CLINICAL TRIAL: NCT02085772
Title: Is Impaired Activation and Migration of Circulating Leukocytes Associated With Overdue Birth in Obese Women?
Brief Title: Leukocytes - ObeSity - Spontaneous Labour
Acronym: LOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: WENDREMAIRE APJ 2013
Record Dates: First submitted 2014-03-05; First posted 2014-03-13 (Estimated); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pre-conceptional Obesity

ARMS (1):
- Patients with pre-conceptional obesity (Experimental)
  Interventions: Other: Blood samples at 37-38 Weeks of amenorrhea; Other: Blood samples at 41 Weeks of amenorrhea if prolonged pregnancy; Other: Blood samples at the time of delivery

INTERVENTIONS:
Other: Blood samples at 37-38 Weeks of amenorrhea
Other: Blood samples at 41 Weeks of amenorrhea if prolonged pregnancy
Other: Blood samples at the time of delivery

SUMMARY:
This is a single-centre observational, prospective study carried out at the maternity unit of Dijon CHU. It will include pregnant women with a pre-conception BMI ≥ 30 kg/m² and will evaluate in these patients, the activation and migration capacities of circulating leukocytes and their association with the onset of spontaneous labour.

Patients who meet the inclusion criteria will be informed about the study during their consultation at the 7th or 8th month, and their gynecologist will invite them to take part. If the answer is positive, the patients will be seen again at a specific consultation for the study between the 37th and 38the Weeks of amenorrhea at the maternity unit of Dijon CHU. During this consultation, the gynecologist will conduct a medical examination, while the Plurithematic clinical investigation center nurse will take a blood sample (3 x 6ml tubes and 1 x 7ml tube).

If labour has not started by 41 Weeks of amenorrhea, the patients will be seen at another consultation (consultation programmed in the usual follow-up of pregnancy) and a second blood sample (1 x 6ml tube and 1 x 7ml) will be taken.

The patients will be followed until childbirth and will be split into two groups according to whether or not they gave birth after the onset of spontaneous labour.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given its written consent
* Please affiliated to a social security scheme
* Body Mass Index Preconception ≥ 30 kg / m²
* Age> 18 years
* Unique Pregnancy
* Having a plot of Normal Fetal heart rate

Exclusion Criteria:

* Pathology changing the mode of delivery or induction of labor (pre-eclampsia, chronic hypertension or gestational, diabetes under unbalanced diet, ...)
* Scheduled Caesarean
* Infectious Disease suspected or proven, including HIV infection, hepatitis C, hepatitis B
* Pathology inflammatory or autoimmune
* Anti-inflammatory or immunosuppressive therapy
* Patient under guardianship
* Patient in safeguarding justice

  • SECONDARY EXCLUSION CRITERIA:
* Caesarean section before labor
* Delivery before 37 Weeks of amenorrhea
* Anti-inflammatory or immunosuppressive therapy during study participation
* Fetal Heart Rate abnormal during study participation
* Premature rupture of fetal membranes without formal labor spontaneously within 48 hours
* Induction of labor or cervical ripening before 41SA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
To determine the initiation of spontaneous labour | Women will be followed until the release of motherhood after giving birth

SECONDARY OUTCOMES:
Occurrence of a vaginal delivery | Women will be followed until the release of motherhood after giving birth
Occurrence of prolonged pregnancy | Women will be followed until the release of motherhood after giving birth
Occurrence of a term exceeding | Women will be followed until the release of motherhood after giving birth

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France